CLINICAL TRIAL: NCT04849533
Title: A Randomized, Multicenter Study of Belatacept, Everolimus, rATG and Early Steroid Withdrawal Versus Belatacept, Mycophenolate, rATG and Chronic Steroids in Renal Transplantation
Brief Title: Belatacept With Early Steroid Withdrawal rATG and Everolimus in Renal Transplantation (BETTER Trial)
Acronym: BETTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Rita Alloway, Professor of Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-423
Record Dates: First submitted 2020-06-29; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Abatacept; Everolimus; Mycophenolic Acid; Adrenal Cortex Hormones; Prednisone; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D Bela/EVR (Experimental): rATG induction/belatacept/everolimus/early steroid withdrawal rATG 1.5mg/kg IV X 4 doses over 10 days belatacept 10mg/kg IV X 1 on POD 1, POD 5, weeks 2, 4, 8, and 12 then 5mg/kg IV X 1 on week 16 and then every 4 weeks thereafter Steroid taper x 5 days (500mg IV, 250mg IV, 125mg IV, 80mg po, 60mg po) Everolimus started within 24hours at 2mg BID and dosed to level 3-8ng/ml
  Interventions: Drug: Belatacept; Drug: Everolimus; Drug: rabbit antithymocyte globulin
- Group E Bela/MMF (Active Comparator): rATG induction/belatacept/mycophenolate/chronic steroidsrATG 1.5mg/kg IV X 4 doses over 10 days belatacept 10mg/kg IV X 1 on POD 1, POD 5, weeks 2, 4, 8, and 12 then 5mg/kg IV X 1 on week 16 and then every 4 weeks thereafter Steroid taper x 5 days (500mg IV, 250mg IV, 125mg IV, 80mg po, 60mg po) and then 5mg po daily thereafter MMF 1gm BID started pre-op and then continued throughout study
  Interventions: Drug: Belatacept; Drug: mycophenolate mofetil; Drug: corticosteroids; Drug: rabbit antithymocyte globulin

INTERVENTIONS:
Drug: Belatacept — belatacept with everolimus is experimental regimen and it is compared to the labeled regimen of belatacept with mycophenolate with steroids for prevention of rejection in renal transplant recipients
  Other Names: Nulojix
Drug: Everolimus — belatacept with everolimus is experimental regimen and it is compared to the labeled regimen of belatacept with mycophenolate with steroids for prevention of rejection in renal transplant recipients
  Other Names: Zortress
  Arms: Group D Bela/EVR
Drug: mycophenolate mofetil — belatacept with mycophenolate is approved regimen for prevention of rejection
  Other Names: Cellcept
  Arms: Group E Bela/MMF
Drug: corticosteroids — belatacept with chronic steroids is approved regimen for prevention of rejection
  Other Names: Prednisone
  Arms: Group E Bela/MMF
Drug: rabbit antithymocyte globulin — rabbit antithymocyte globulin induction for prevention of rejection
  Other Names: rATG, thymoglobulin

SUMMARY:
This study is designed to determine the safety and efficacy of two calcineurin inhibitor free treatment groups 1) a belatacept, everolimus and early corticosteroid withdrawal (ECSWD) immunosuppressive regimen with rabbit antithymocyte globulin induction (rATG) and 2) a belatacept, mycophenolate, chronic steroid regimen with rATG and compare to historical controls of tacrolimus-based and belatacept-based regimens in combination with rATG induction, mycophenolate, and ESWD in renal transplant recipients.

The purpose is to evaluate the effect of 2 regimens (rATG induction/belatacept/everolimus/ESWD and rATG induction/belatacept/mycophenolate/CS) on the composite of patient death, graft loss, or eGFR (MDRD) < 45 mL/min/1.73m2 at Month 12 post-transplantation compared to historical controls of the BEST Trial (groups B and C).

DETAILED DESCRIPTION:
The BETTER trial is designed to determine the safety and efficacy of two calcineurin inhibitor free treatment groups 1) a belatacept, everolimus and early corticosteroid withdrawal (ESWD) immunosuppressive regimen with rabbit antithymocyte globulin induction (rATG) and 2) a belatacept, mycophenolate, chronic steroid regimen with rATG and compare to historical controls of tacrolimus-based and belatacept-based regimens in combination with rATG induction, mycophenolate, and ESWD in renal transplant recipients.

Study Hypotheses

1. A belatacept-based immunosuppressive regimen with rATG induction, everolimus and ESWD in renal transplant recipients will lead to less risk of graft loss, patient death, or eGFR <45ml/min/1.73m2 at 12 and 24 months as compared to a tacrolimus-based immunosuppressive regimen with rATG, mycophenolate, and ESWD in renal transplant recipients (historical control from the BEST Trial-Group C).
2. A belatacept-based immunosuppressive regimen with rATG induction, everolimus and ESWD in renal transplant recipients will lead to less risk of graft loss, patient death, or eGFR <45ml/min/1.73m2 at 12 and 24 months as compared to a belatacept-based immunosuppressive regimen with rATG and mycophenolate, and ESWD in renal transplant recipients (historical control from the BEST Trial-Group B).
3. A belatacept-based immunosuppressive regimen with rATG, mycophenolate and CS in renal transplant recipients will lead to less risk of graft loss, patient death, or eGFR <45ml/min/1.73m2 at 12 and 24 months as compared to a tacrolimus-based immunosuppressive regimen with rATG, mycophenolate, and ESWD in renal transplant recipients (historical control from the BEST Trial-Group C).
4. A belatacept-based immunosuppressive regimen with rATG induction, mycophenolate and CS in renal transplant recipients will lead to less risk of graft loss, patient death, or eGFR <45ml/min/1.73m2 at 12 and 24 months as compared to a belatacept-based immunosuppressive regimen with rATG, mycophenolate, and ESWD in renal transplant recipients (historical control from the BEST Trial-Group B).

A controlled, randomized group study is accepted in renal transplantation to evaluate new immunosuppressive regimens versus the current standard of care. Although the ideal study would employ a blinded methodology with a simultaneous control group to minimize bias, the study will not be blinded and evaluates a historical control groups conducted in similar centers.

To allow comparison between studies, the primary composite endpoint of death, graft loss, or eGFR <45ml/min/1.73m2 will be analyzed similarly. The secondary and tertiary endpoints are the similar as well.

The BETTER study proposes to compare two additional treatment groups of rATG/belatacept/everolimus/ESWD (Group D) and rATG/belatacept/mycophenolate/CS (Group E) to the historical control Groups B and C.

All immunosuppressive agents are approved by the FDA for the prophylaxis of renal transplant rejection, and will be dosed and administered consistent with current clinical practice.

ELIGIBILITY:
Inclusion criteria

1. Male and female patients ≥ 18 years of age.
2. Patient who is receiving a renal transplant from a living or heart-beating deceased donor.
3. Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to study inclusion.
4. The patient has given written informed consent to participate in the study

Exclusion criteria

1. Patient has previously received an organ transplant other than a kidney.
2. Patient is receiving an HLA identical living donor transplant.
3. Patient who is a recipient of a multiple organ transplant.
4. Patient has a most recent cytotoxic PRA of >25% or calculated PRA >50% where multiple moderate level HLA antibodies exist and in the opinion of the PI represents substantial HLA sensitization.
5. Patient with a positive T or B cell crossmatch that is primarily due to HLA antibodies.
6. Patient with a donor specific antibody (DSA) as deemed by the PI to be associated with significant risk of rejection.
7. Patient has received an ABO incompatible donor kidney.
8. The deceased donor and/or deceased donor kidney meet any of the following extended criteria for organ donation (ECD):

   1. Donor age ≥ 60 years OR
   2. Donor age 50-59 years and 1 of the following:

   i. Cerebrovascular accident (CVA) + hypertension + SCr > 1.5 mg/dL OR ii. CVA + hypertension OR iii. CVA + SCr > 1.5 mg/dL OR iv. Hypertension + SCr > 1.5 mg/dL OR c. CIT ≥ 24 hours, donor age > 10 years OR d. Donation after cardiac death (DCD)
9. Recipients will be receiving a dual or en bloc kidney transplant.
10. Donor anticipated cold ischemia is > 30 hours.
11. Recipient that is seropositive for hepatitis C virus (HCV) with detectable Hepatitis C viral load are excluded. HCV seropositive patients with a negative HCV viral load testing may be included.
12. Recipients receiving a kidney from a donor with HCV viremia (detected through nucleic acid testing or other means)
13. Recipients with a positive hepatitis B viral load or positive hepatitis B surface antigen testing within 1 year of consent.
14. Hepatitis B surface antibody negative recipients receiving a kidney from a donor seropositive for hepatitis B core antibody or hepatitis B nucleic acid.
15. Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
16. Recipient who is seronegative for Epstein Barr Virus (EBV)
17. Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
18. Patients with thrombocytopenia (PLT <75,000/mm3), and/or leukopenia (WBC < 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
19. Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
20. Patient who has undergone desensitization therapy within 6 months prior to transplant.
21. Patient has a known hypersensitivity to belatacept, tacrolimus, mycophenolate mofetil/mycophenolic acid, everolimus, rabbit anti-thymocyte globulin, or glucocorticoids.
22. Patient is receiving chronic steroid therapy at the time of transplant.
23. Patients with a history of cancer (other than non-melanoma skin cell cancers cured by local resection) within the last 5 years, unless they have an expected disease-free survival of >95%.
24. Patient is pregnant, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
25. Women of childbearing potential must use reliable contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
26. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
27. Inability to cooperate or communicate with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of patient death, graft loss, or eGFR (MDRD) < 45ml/min mL/min/1.73m2 | 12 months
  Number of subjects with composite endpoint of either patient death, graft loss, or eGFR (MDRD) < 45 mL/min/1.73m2 at Month 12 post-transplantation compared to historical controls of the BEST Trial (groups B and C).

SECONDARY OUTCOMES:
Incidence of Biopsy-proven acute rejection (BPAR) by Banff 2007 criteria stratified by type (ACR, AMR, or Mixed rejection) | 12 and 24 months
  To evaluate, by treatment group at 12 and 24 months incidence of various rejection types
Incidence of graft survival censored by patients who died with functioning graft | 12 and 24 months
  Incidence of death-censored graft survival not including any patients who died with their graft still functioning
# of Patients with eGFR (MDRD) < 30 mL/min/1.73m2 | 12 and 24 months
  # of subjects with eGFR (MDRD) < 30 mL/min/1.73m2
# Patients with development of de novo donor specific antibody (DSA) | 12 and 24 months
  Patients with development of de novo donor specific antibody (DSA) after transplant
Composite endpoint of patient death, graft loss, or estimated eGFR (MDRD) < 45 mL/min/1.73m2 at Month 24 post-transplantation | 24 months
  Composite endpoint of patients with either death, graft loss, or estimated eGFR (MDRD) < 45 mL/min/1.73m2 at Month 24 post-transplantation
# Patients with Incidence of Infections | 12 and 24 months
  Incidence of infections, including CMV and BK virus

CONTACTS AND LOCATIONS:
Overall Officials: Rita R Alloway, PharmD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No